CLINICAL TRIAL: NCT02493868
Title: A Randomized, Double-blind, Multicenter, Active-Controlled Study of Intranasal Esketamine Plus an Oral Antidepressant for Relapse Prevention in Treatment-resistant Depression
Brief Title: A Study of Intranasal Esketamine Plus an Oral Antidepressant for Relapse Prevention in Adult Participants With Treatment-resistant Depression
Acronym: SUSTAIN-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR107128; ESKETINTRD3003 (Other: Janssen Research & Development, LLC); 2014-004586-24 (EudraCT Number)
Record Dates: First submitted 2015-05-13; First posted 2015-07-10 (Estimated); Results first posted 2019-05-21 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Depressive Disorder, Treatment-Resistant
Keywords: Treatment-resistant Depression; Esketamine; Placebo; Oral Antidepressant; Relapse prevention
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Esketamine; Duloxetine Hydrochloride; Antidepressive Agents; Escitalopram; Sertraline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Intranasal Esketamine plus oral antidepressant (Experimental): Open-Label Induction Phase: Direct-entry participants will self-administer esketamine intranasally twice per week for 4 weeks as a flexible dose regimen in the Open-label Induction Phase. Participants will initiate a new oral antidepressant on Day 1 of this phase. Optimization Phase: Direct-entry and transferred-entry participants will self-administer intranasal esketamine (same dose) at weekly treatment sessions for the first 4 weeks of this phase, then individualized to either once weekly or once every other week based on depressive symptoms. Participants continue same oral antidepressant treatment from induction phase. Maintenance Phase: Direct-entry and transferred-entry participants assigned to esketamine will self-administer intranasal esketamine (same dose) once weekly or once every other week based on depressive symptoms. Participants continue same oral antidepressant treatment from induction phase.
  Interventions: Drug: Esketamine; Drug: Duloxetine (Oral Antidepressant); Drug: Escitalopram (Oral antidepressant); Drug: Sertraline (Oral Antidepressant); Drug: Venlafaxine Extended Release (XR) (Oral Antidepressant)
- Placebo Plus Oral Antidepressant (Experimental): Optimization Phase: Transferred-entry participants will self-administer intranasal placebo at weekly treatment sessions for the first 4 weeks of this phase, then individualized to either once weekly or once every other week based on depressive symptoms. Participants continue same oral antidepressant treatment from induction phase. Maintenance Phase: Direct-entry and transferred-entry participants assigned to intranasal placebo will self-administer intranasal placebo once weekly or once every other week based on depressive symptoms. Participants continue same oral antidepressant treatment from induction phase.
  Interventions: Drug: Placebo; Drug: Duloxetine (Oral Antidepressant); Drug: Escitalopram (Oral antidepressant); Drug: Sertraline (Oral Antidepressant); Drug: Venlafaxine Extended Release (XR) (Oral Antidepressant)

INTERVENTIONS:
Drug: Esketamine — Open-label induction phase: Direct entry participants start at a dose of 56 mg on Day 1. On Day 4, the dose may be increased to 84 mg or remain at 56 mg. From Day 8 to 22, dose may be increased to 84 mg, remain the same or be reduced to 56 mg from 84 mg per protocol, at investigator's discretion based on efficacy and/or tolerability. On Day 25, a dose reduction from 84 mg to 56 mg is permitted but no dose increase is permitted. Optimization Phase: Direct-entry and transferred-entry participants will self-administer intranasal esketamine (same dose) for first 4 weeks, then individualized to either once weekly or once every other week based on depressive symptoms. Maintenance Phase: All participants assigned to esketamine will self-administer intranasal esketamine once weekly or once every other week based on depressive symptoms.
  Arms: Intranasal Esketamine plus oral antidepressant
Drug: Placebo — Optimization Phase: Transferred-entry participant will self-administer intranasal placebo at weekly treatment sessions for the first 4 weeks of this phase, then individualized to either once weekly or once every other week based on depressive symptoms. Maintenance Phase: Direct-entry and transferred-entry participants assigned to placebo will self-administer matching intranasal placebo once weekly or once based on depressive symptoms.
  Arms: Placebo Plus Oral Antidepressant
Drug: Duloxetine (Oral Antidepressant) — Duloxetine could be selected as the oral antidepressant medication by the investigator based on review of Massachusetts General Hospital - Antidepressant Treatment Response Questionnaire (MGH-ATRQ) and relevant prior antidepressant medication information. The minimum therapeutic dose is 60 milligram per day (mg/day).
Drug: Escitalopram (Oral antidepressant) — Escitalopram could be selected as the oral antidepressant medication by the investigator based on review of MGH-ATRQ and relevant prior antidepressant medication information. Escitalopram will be titrated upto a maximum dose of 20 mg/day, but if not tolerated the dose can be reduced to the minimum therapeutic dose of 10 mg/day.
Drug: Sertraline (Oral Antidepressant) — Sertraline could be selected as the oral antidepressant medication by the investigator based on review of MGH-ATRQ and relevant prior antidepressant medication information. Sertraline will be titrated upto a maximum dose of 200 mg/day, but if not tolerated the dose can be reduced to the minimum therapeutic dose of 50 mg/day.
Drug: Venlafaxine Extended Release (XR) (Oral Antidepressant) — Venlafaxine Extended Release could be selected as the oral antidepressant medication by the investigator based on review of MGH-ATRQ and relevant prior antidepressant medication information. Venlafaxine Extended Release will be titrated upto a maximum dose of 225 mg/day, but if not tolerated the dose can be reduced to the minimum therapeutic dose of 150 mg/day.

SUMMARY:
The purpose of this study is to assess the efficacy of intranasal esketamine plus an oral antidepressant compared with an oral antidepressant (active comparator) plus intranasal placebo in delaying relapse of depressive symptoms in participants with treatment-resistant depression (TRD) who are in stable remission after an induction and optimization course of intranasal esketamine plus an oral antidepressant.

DETAILED DESCRIPTION:
This is a randomized, double-blind (neither the researchers nor the participant know what treatment the participants is receiving), active-controlled, multicenter (more than 1 study site) study in participants with TRD to assess the efficacy of intranasal esketamine plus an oral antidepressant compared with an oral antidepressant (active comparator) plus intranasal placebo in delaying relapse of depressive symptoms. The study will consist of 5 phases: Screening/Prospective Observational Phase (4-7weeks) for direct-entry participants only, Open-label Induction Phase (4-weeks) for direct-entry participants only, Optimization Phase (12-weeks; open-label for direct-entry participants and double-blind for transferred-entry participants), Maintenance Phase (variable duration; double-blind for all participants) and Follow-up Phase (2-weeks). Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

For Direct-Entry Participants

* At the time of signing the informed consent form (ICF), participant must be a man or woman 18 (or older if the minimum legal age of consent in the country in which the study is taking place is greater than [>]18) to 64 years of age, inclusive - At the start of the screening/prospective observational phase, participant must meet the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) diagnostic criteria for single-episode major depressive disorder (MDD) (if single-episode MDD, the duration must be greater than or equal to [>=] 2 years) or recurrent MDD, without psychotic features, based upon clinical assessment and confirmed by the Mini-International Neuropsychiatric Interview (MINI)
* At the start of the screening/prospective observational phase, participant must have an Inventory of Depressive Symptomatology-Clinician rated ( IDS-C30) total score of greater than or equal to (>=) 34
* At the start of the screening/prospective observational phase, participants must have had nonresponse (less than or equal to 25 percent [%] improvement) to greater than or equal to (>=1) but less than or equal to (<=) 5 oral antidepressant treatments taken at adequate dosage and for adequate duration, as assessed using the Massachusetts General Hospital (MGH-ATRQ )
* MGH-ATRQ and documented by medical history and pharmacy/prescription records, for the current episode of depression. In addition, the participant is taking different ongoing oral antidepressant treatment (on the MGH-ATRQ) for at least the previous 2 weeks at or above the minimal therapeutic dose
* The participant's current major depressive episode, depression symptom severity (Week 1 MADRS total score >=28 required), and treatment response to antidepressant treatments used in the current depressive episode (retrospectively assessed) must be deemed valid for participation in a clinical study based on a Site-Independent Qualification Assessment For Transferred-Entry Participants
* The participant must have completed the double-blind induction phase in ESKETINTRD3001 or ESKETINTRD3002 and must have demonstrated response at the end of that phase (>=50% reduction in the MADRS total score from baseline [Day 1 pre-randomization] at the end of the 4-week double-blind induction phase)

Exclusion Criteria:

* Participants who have previously demonstrated nonresponse of depressive symptoms to esketamine or ketamine in the current major depressive episode, to all 4 of the oral antidepressant treatment options available for the double-blind induction phase (ie, duloxetine, escitalopram, sertraline, and venlafaxine extended release [XR]) in the current major depressive episode (based on MGH-ATRQ), or an adequate course of treatment with electroconvulsive therapy (ECT) in the current major depressive episode, defined as at least 7 treatments with unilateral/bilateral ECT
* Participant has received vagal nerve stimulation (VNS) or has received deep brain stimulation (DBS) in the current episode of depression
* Participant has a current or prior DSM-5 diagnosis of a psychotic disorder or MDD with psychotic features, bipolar or related disorders (confirmed by the MINI), obsessive compulsive disorder (current only), intellectual disability (DSM-5 diagnostic codes 317, 318.0, 318.1, 318.2, 315.8, and 319), autism spectrum disorder, borderline personality disorder, antisocial personality disorder, histrionic personality disorder, or narcissistic personality disorder
* Participant has homicidal ideation/intent, per the investigator's clinical judgment, or has suicidal ideation with some intent to act within 6 months prior to the start of the screening/prospective observational phase, per the investigator's clinical judgment or based on the Columbia Suicide Severity Rating Scale (C-SSRS)
* Participants with history of moderate or severe substance or alcohol use disorder according to DSM-5 criteria

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 719 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (155):
- United States (53):
  - Birmingham, Alabama
  - Little Rock, Arkansas
  - Anaheim, California
  - Garden Grove, California
  - Glendale, California
  - Oakland, California
  - Orange, California
  - San Diego, California
  - San Marcos, California
  - San Rafael, California
  - Hartford, Connecticut
  - Bradenton, Florida
  - Gainesville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Hoffman Estates, Illinois
  - Joliet, Illinois
  - Maywood, Illinois
  - Schaumburg, Illinois
  - Skokie, Illinois
  - Prairie Village, Kansas
  - Wichita, Kansas
  - Lake Charles, Louisiana
  - Baltimore, Maryland
  - Gaithersburg, Maryland
  - Boston, Massachusetts
  - New Bedford, Massachusetts
  - Quincy, Massachusetts
  - Watertown, Massachusetts
  - Worcester, Massachusetts
  - Rochester Hills, Michigan
  - Minneapolis, Minnesota
  - O'Fallon, Missouri
  - Saint Charles, Missouri
  - Omaha, Nebraska
  - New York, New York
  - Durham, North Carolina
  - Hickory, North Carolina
  - Oklahoma City, Oklahoma
  - Media, Pennsylvania
  - Philadelphia, Pennsylvania
  - Scranton, Pennsylvania
  - Lincoln, Rhode Island
  - Providence, Rhode Island
  - Arlington, Texas
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - Charlottesville, Virginia
  - Waukesha, Wisconsin
- Belgium (6):
  - Aalst
  - Bruges
  - Brussels
  - Heusden-Zolder
  - Liège
  - Yvoir
- Brazil (11):
  - Belo Horizonte
  - Curitiba
  - Fortaleza
  - Goiânia
  - Itapira
  - Passo Fundo
  - Porto Alegre
  - Rio de Janeiro
  - Santo André
  - São José do Rio Preto
  - São Paulo
- Canada (6):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Kingston, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Czechia (8):
  - Brno
  - Hostivice
  - Klecany
  - Kutná Hora
  - Litoměřice
  - Pilsen
  - Prague
  - Strakonice
- Estonia (3):
  - Pärnu
  - Tallinn
  - Tartu
- France (7):
  - Clermont-Ferrand
  - Douai
  - Nantes
  - Nîmes
  - Paris
  - Poitiers
  - Toulon
- Germany (8):
  - Berlin
  - Cham
  - Gelsenkirchen
  - Halle
  - Mainz
  - Mittweida
  - Pfaffenhofen
  - Prien am Chiemsee
- Hungary (9):
  - Balassagyarmat
  - Budapest
  - Debrecen
  - Győr
  - Pécs
  - Sopron
  - Szeged
  - Szekszárd
  - Vác
- Mexico (5):
  - Guadalajara
  - León
  - Mexico City
  - Monterrey
  - San Luis Potosí City
- Poland (11):
  - Bełchatów
  - Bialystok
  - Bydgoszcz
  - Gdansk
  - Leszno
  - Lodz
  - Lublin
  - Pruszków
  - Torun
  - Tuszyn
  - Warsaw
- Slovakia (5):
  - Bratislava
  - Liptovský Mikuláš
  - Rimavská Sobota
  - Rožňava
  - Svidník
- Spain (8):
  - Alcorcón
  - Barcelona
  - Palma
  - Pamplona
  - Ponferrada
  - Sabadell
  - Salamanca
  - Vitoria-Gasteiz
- Sweden (4):
  - Lund
  - Skövde
  - Solna
  - Stockholm
- Turkey (Türkiye) (11):
  - Adana
  - Ankara
  - Bursa
  - Denizli
  - Istanbul
  - Izmir
  - Kucukcekmece/Istanbul
  - Manisa
  - Oanakkale
  - Sakarya
  - Samsun

REFERENCES:
- [Derived] Kern Sliwa J, Naranjo RR Jr, Turkoz I, Petrillo MP, Cabrera P, Trivedi M. Effects of esketamine nasal spray on depressive symptom severity in adults with treatment-resistant depression and associations between the Montgomery-Asberg Depression Rating Scale and the 9-item Patient Health Questionnaire. CNS Spectr. 2024 Jun;29(3):176-186. doi: 10.1017/S1092852924000105. Epub 2024 Apr 1. PMID 38557430
- [Derived] Castro M, Wilkinson ST, Al Jurdi RK, Petrillo MP, Zaki N, Borentain S, Fu DJ, Turkoz I, Sun L, Brown B, Cabrera P. Efficacy and Safety of Esketamine Nasal Spray in Patients with Treatment-Resistant Depression Who Completed a Second Induction Period: Analysis of the Ongoing SUSTAIN-3 Study. CNS Drugs. 2023 Aug;37(8):715-723. doi: 10.1007/s40263-023-01026-3. Epub 2023 Aug 9. PMID 37558912
- [Derived] Williamson DJ, Gogate JP, Kern Sliwa JK, Manera LS, Preskorn SH, Winokur A, Starr HL, Daly EJ. Longitudinal Course of Adverse Events With Esketamine Nasal Spray: A Post Hoc Analysis of Pooled Data From Phase 3 Trials in Patients With Treatment-Resistant Depression. J Clin Psychiatry. 2022 Sep 19;83(6):21m14318. doi: 10.4088/JCP.21m14318. PMID 36149841
- [Derived] Chen G, Chen L, Zhang Y, Li X, Lane R, Lim P, Daly EJ, Furey ML, Fedgchin M, Popova V, Singh JB, Drevets WC. Relationship Between Dissociation and Antidepressant Effects of Esketamine Nasal Spray in Patients With Treatment-Resistant Depression. Int J Neuropsychopharmacol. 2022 Apr 19;25(4):269-279. doi: 10.1093/ijnp/pyab084. PMID 35022754
- [Derived] Doty RL, Popova V, Wylie C, Fedgchin M, Daly E, Janik A, Ochs-Ross R, Lane R, Lim P, Cooper K, Melkote R, Jamieson C, Singh J, Drevets WC. Effect of Esketamine Nasal Spray on Olfactory Function and Nasal Tolerability in Patients with Treatment-Resistant Depression: Results from Four Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase III Studies. CNS Drugs. 2021 Jul;35(7):781-794. doi: 10.1007/s40263-021-00826-9. Epub 2021 Jul 7. PMID 34235612
- [Derived] Katz EG, Hough D, Doherty T, Lane R, Singh J, Levitan B. Benefit-Risk Assessment of Esketamine Nasal Spray vs. Placebo in Treatment-Resistant Depression. Clin Pharmacol Ther. 2021 Feb;109(2):536-546. doi: 10.1002/cpt.2024. Epub 2020 Oct 13. PMID 32860422
- [Derived] Daly EJ, Trivedi MH, Janik A, Li H, Zhang Y, Li X, Lane R, Lim P, Duca AR, Hough D, Thase ME, Zajecka J, Winokur A, Divacka I, Fagiolini A, Cubala WJ, Bitter I, Blier P, Shelton RC, Molero P, Manji H, Drevets WC, Singh JB. Efficacy of Esketamine Nasal Spray Plus Oral Antidepressant Treatment for Relapse Prevention in Patients With Treatment-Resistant Depression: A Randomized Clinical Trial. JAMA Psychiatry. 2019 Sep 1;76(9):893-903. doi: 10.1001/jamapsychiatry.2019.1189. PMID 31166571
- See also: A Randomized, Double-blind, Multicenter, Active-controlled Study of Intranasal Esketamine Plus an Oral Antidepressant for Relapse Prevention in Treatment-resistant Depression — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR107128&attachmentIdentifier=d913e5fa-3636-4665-a11c-7b69d8a8df62&fileName=ESKETINTRD3003_(CR107128)_Additional_results_data_CH.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total of 719 participants were enrolled out of which 705 were included in the analysis. 14 participants were excluded due to premature closure of a site due to quality and data integrity issues.
Pre-assignment Details: Out of 705 participants, 437 (direct entry [DE] participants) entered in induction (IND) phase and 268 participants (150 transferred-entry [TE] participants from study ESKETINTRD3001 [NCT02417064] and 118 participants from study ESKETINTRD3002 [NCT02418585]) entered in this study in optimization (OP) phase.
Groups:
- Intranasal Esketamine + Oral AD: Open-label induction (IND) phase (DE): received 56 or 84 milligram intranasal esketamine solution twice weekly with open-label oral AD (one of: duloxetine/escitalopram/sertraline/venlafaxine extended release [XR]), once daily for 4 weeks. OP phase (DE+TE): received intranasal esketamine (same dose) solution once per week for first 4 weeks, then once per week/once every other week based on severity of depressive symptoms, and continued same oral AD from IND phase for 12 weeks. MA phase (DE+TE): Participants were randomized (at end of OP phase) to receive intranasal esketamine (same dose) once weekly/once every other week based on depressive symptoms and continued same oral AD from IND phase. Follow-up (FU) phase: participants received no intranasal esketamine but continued oral AD for 2 weeks unless determined to not be clinically appropriate. Participants who were non-responders at end of IND phase or who were early terminated at any phase proceeded directly to FU phase.
- Oral AD + Intranasal Placebo: Open-label induction phase: No intervention was administered. Optimization phase (transferred-entry participants): received intranasal esketamine matching placebo solution once per week for the first 4 weeks, then once per week or once every other week depending on severity of depressive symptoms with open-label oral antidepressant (AD) (one of: duloxetine/escitalopram/sertraline/venlafaxine XR), once daily for 12 weeks. Maintenance (MA) phase (DE+TE participants): Participants were randomized (at the end of optimization phase) to receive intranasal esketamine placebo with oral AD from optimization phase. Follow-up Phase: participants received oral AD for 2 weeks of the follow-up phase unless it was determined to not be clinically appropriate. Participants who were non-responders at end of IND phase or who were early terminated at any phase proceeded directly to FU phase.
Period: Induction Phase: DE Participants
Arm/Group | Intranasal Esketamine + Oral AD | Oral AD + Intranasal Placebo
Started | 437 | 0
Completed | 273 (Participants who completed and met predefined response criteria continued to OP phase.) | 0
Not Completed | 164 | 0
Not completed — Adverse Event | 22 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Lack of Efficacy | 2 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 15 | 0
Not completed — Not meet criteria to continue next phase | 114 | 0
Not completed — Other | 8 | 0
Period: Optimization Phase: DE+TE Participants
Arm/Group | Intranasal Esketamine + Oral AD | Oral AD + Intranasal Placebo
Started | 455 (Total participants: direct-entry (273) + esketamine-treated transferred-entry participants (182).) | 86 (Placebo treated transferred-entry participant.)
Completed | 297 (Participants who completed and met predefined remission/response criteria randomized to MA phase) | 54 (Participants who completed and met predefined remission/response criteria continued to MA phase.)
Not Completed | 158 | 32
Not completed — Adverse Event | 5 | 0
Not completed — Lost to Follow-up | 2 | 1
Not completed — Lack of Efficacy | 8 | 0
Not completed — Protocol Violation | 4 | 1
Not completed — Withdrawal by Subject | 8 | 3
Not completed — MADRS >= 22 for 2 Consecutive Visit | 14 | 5
Not completed — Not meet criteria to continue next phase | 107 | 20
Not completed — Other | 10 | 2
Period: Maintenance Phase: DE+TE Participants
Arm/Group | Intranasal Esketamine + Oral AD | Oral AD + Intranasal Placebo
Started | 152 (152 participants randomized from intranasal esketamine arm after OP phase: DE (90) + TE (62)) | 199 (145 participants randomized from intranasal esketamine arm after OP phase+54 continued from OP phase)
Stable Remitters | 90 | 86
Stable Responders | 62 | 59
Completed | 139 | 177
Not Completed | 13 | 22
Not completed — Adverse Event | 1 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 5 | 7
Not completed — Pregnancy | 1 | 0
Not completed — Non Compliance with Study Drug | 0 | 1
Not completed — Other | 4 | 9
Period: Follow-up Phase
Arm/Group | Intranasal Esketamine + Oral AD | Oral AD + Intranasal Placebo
Started | 481 | 64
Completed | 470 | 62
Not Completed | 11 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Investigator Decision | 5 | 1
Not completed — Other | 2 | 1

BASELINE CHARACTERISTICS:
Population: The baseline characteristics are reported for the all enrolled population. Not all participants enrolled were actually randomized to one of 2 treatments in the Maintenance phase as they had to meet specific criteria to be randomized.
Groups:
- All Participants: All Participants (direct entry and transferred entry) who were enrolled in this study and received intranasal esketamine, matching placebo and oral antidepressant as per the assigned treatment.
Arm/Group | All Participants
Number analyzed (Participants) | 705
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 457
  Male | 248
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 94
  Not Hispanic or Latino | 600
  Unknown or Not Reported | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3
  Black or African American | 31
  Hispanic or Latino | 71
  Other | 38
  White Non-Hispanic | 562
Region of Enrollment [Count of Participants; unit: Participants]
  BELGIUM | 14
  BRAZIL | 64
  CANADA | 5
  CZECH REPUBLIC | 99
  ESTONIA | 1
  FRANCE | 10
  GERMANY | 7
  HUNGARY | 35
  ITALY | 21
  MEXICO | 35
  POLAND | 132
  SLOVAKIA | 7
  SPAIN | 16
  SWEDEN | 16
  TURKEY | 53
  UNITED STATES | 190

OUTCOME MEASURES:

1. Primary Outcome: Time to Relapse in Participants With Stable Remission (Maintenance Phase)
Description: Relapse is defined as any of following: Montgomery-asberg depression rating scale (MADRS) total score greater than or equal to (>=) 22 for 2 consecutive assessments separated by 5-15 days and/or hospitalization for worsening depression or any other clinically relevant event to be suggestive of a relapse of depressive illness such as suicide attempt/completed suicide/hospitalization for suicide prevention; If hospitalized, start date of hospitalization will be date of relapse, if not hospitalized date of event will be used. MADRS: clinician-rated scale to measure depression severity and to detect changes due to antidepressant treatment. It has 10 items, scored from 0-6 (not present/normal-severe/continuous symptoms), with total score of 60. Higher scores mean more severe condition. Stable remission: MADRS total score less than or equal to (<=) 12 for at least 3 of last 4 weeks of OP phase, with 1 excursion total score greater than (>) 12 or one missing assessment at OP week 13 or 14.
Time Frame: Time from randomization to the first relapse during the maintenance phase (up to 92 Weeks)
Population: Full (stable remitters) analysis set included all the randomized participants who were in stable remission at the end of the optimization phase and received at least 1 dose of intranasal study drug and 1 dose of oral AD during the maintenance phase.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Oral AD+ Intranasal Placebo: Open-label induction phase: No intervention was administered. Optimization phase (transferred-entry participants): received intranasal esketamine matching placebo solution once per week for the first 4 weeks, then once per week or once every other week depending on severity of depressive symptoms with open-label oral antidepressant (AD) (one of: duloxetine/escitalopram/sertraline/venlafaxine XR), once daily for 12 weeks. Maintenance phase (DE+TE participants): Participants were randomized (at the end of optimization phase) to receive intranasal esketamine placebo with oral AD from optimization phase. Follow-up Phase: Participants received oral AD for 2 weeks of the follow-up phase unless it was determined to not be clinically appropriate. Participants who were non-responders at end of IND phase or who were early terminated at any phase proceeded directly to FU phase.
Arm/Group | Intranasal Esketamine + Oral AD | Oral AD+ Intranasal Placebo
Number analyzed (Participants) | 90 | 86
Days | NA [NA to NA] — Here NA signifies that median and 95%CI was not estimable due to not having sufficient events to meet the threshold for 50% on the Kaplan-Meier curve. | 273.0 [97.0 to NA] — Here NA signifies that upper limit of CI could not be estimated due to insufficient data.
Statistical Analysis 1: Comparison: Intranasal Esketamine + Oral AD vs Oral AD+ Intranasal Placebo; Test type: Superiority; p = 0.003, Weighted Log-rank; Hazard Ratio (HR) = 0.49, 95% CI 2-sided [0.29 to 0.84]

2. Secondary Outcome: Time to Relapse in Participants With Stable Response (But Not in Stable Remission) (Maintenance Phase)
Description: Relapse is defined as any of following: MADRS total score >= 22 for 2 consecutive assessments separated by 5-15 days and/or hospitalization for worsening depression or any other clinically relevant event to be suggestive of a relapse of depressive illness such as suicide attempt/completed suicide/hospitalization for suicide prevention; If hospitalized, start date of hospitalization will be date of relapse, if not hospitalized date of event will be used. MADRS: clinician-rated scale to measure depression severity and to detect changes due to antidepressant treatment. It has 10 items, scored from 0-6 (not present/normal-severe/continuous symptoms), with total score of 60. Higher scores mean more severe condition. Stable response is defined as >= 50 percent (%) reduction in MADRS total score from baseline (Day 1 of induction phase, prior to first intranasal dose) in each of the last 2 weeks of the OP phase, but without meeting criteria for stable remission.
Time Frame: Time from randomization to the first relapse during the maintenance phase (up to 92 Weeks)
Population: Full (stable responders) analysis set included all randomized participants who were stable responders (who were not stable remitters) at the end of the optimization phase and who received at least 1 dose of intranasal study drug and 1 dose of oral antidepressant during the maintenance phase.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Intranasal Esketamine + Oral AD | Oral AD+ Intranasal Placebo
Number analyzed (Participants) | 62 | 59
Days | 635.0 [264.0 to 635.0] | 88.0 [46.0 to 196.0]

3. Secondary Outcome: Change From Baseline in MADRS Total Score at Endpoint in Participants With Stable Remission (Maintenance Phase)
Description: MADRS: clinician-rated scale to measure depression severity and to detect changes due to antidepressant treatment. It has 10 items, scored from 0-6 (not present/normal - severe/continuous symptoms), with total score of 60. Higher scores mean more severe condition. The change from baseline in MADRS total score (last observation carried forward [LOCF] data), at endpoint was reported. The last post baseline observation was carried forward as the endpoint.
Time Frame: Baseline and Endpoint (Up to 92 Weeks)
Population: Full (stable remitters) analysis set included all randomized participants who were in stable remission at end of OP phase and received at least 1 dose of intranasal study drug and 1 dose of oral AD during MA phase. Here 'N' (overall number of participants analyzed) signifies number of participants who were evaluable for this outcome measure (OM).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine + Oral AD | Oral AD+ Intranasal Placebo
Number analyzed (Participants) | 89 | 86
Units on a scale | 7.5 (11.59) | 12.5 (13.63)

4. Secondary Outcome: Change From Baseline in MADRS Total Score at Endpoint in Participants With Stable Response (But Not in Stable Remission) (Maintenance Phase)
Description: MADRS: clinician-rated scale to measure depression severity and to detect changes due to antidepressant treatment. It has 10 items, scored from 0-6 (not present/normal - severe/continuous symptoms), with total score of 60. Higher scores mean more severe condition. The change from baseline in MADRS total score (LOCF data), at endpoint was reported. The last post baseline observation was carried forward as the endpoint.
Time Frame: Baseline and Endpoint (Up to 92 Weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine + Oral AD | Oral AD+ Intranasal Placebo
Number analyzed (Participants) | 62 | 59
Units on a scale | 4.4 (11.38) | 11.4 (12.00)

5. Secondary Outcome: Change From Baseline in Patient Health Questionnaire-9 (PHQ-9) Total Score at Endpoint in Participants With Stable Remission (Maintenance Phase)
Description: PHQ-9 is a 9-item, self-report scale assessing depressive symptoms. Each item is rated on a 4-point scale (0 = Not at all, 1 = Several Days, 2 = More than half the days, and 3 = Nearly every day). The participant's item responses are summed to provide a total score (range of 0 to 27) with higher scores indicating greater severity of depressive symptoms. The severity of the PHQ-9 is categorized as follows: None-minimal (0-4), mild (5-9), moderate (10-14), moderately severe (15-19) and severe (20-27). The change from baseline in PHQ-9 total score, (LOCF data) at endpoint was reported. The last post baseline observation was carried forward as the endpoint.
Time Frame: Baseline and Endpoint (Up to 92 Weeks)
Population: Full (stable remitters) analysis set included all randomized participants who were in stable remission at the end of OP phase and received at least 1 dose of intranasal study drug and 1 dose of oral AD during MA phase. Here 'N' (overall number of participants analyzed) signifies number of participants who were evaluable for this OM.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine + Oral AD | Oral AD+ Intranasal Placebo
Number analyzed (Participants) | 89 | 86
Units on a scale | 3.3 (5.58) | 5.9 (7.09)

6. Secondary Outcome: Change From Baseline in PHQ-9 Total Score at Endpoint in Participants With Stable Response (But Not in Stable Remission) (Maintenance Phase)
Description: as for outcome 5
Time Frame: Baseline and Endpoint (Up to 92 Weeks)
Population: Full (stable responders) analysis set: all randomized participants who were stable responders (not stable remitters) at end of OP phase and received at least 1 dose of intranasal study drug and 1 dose of oral AD during MA phase. Here 'N' (overall number of participants analyzed) signifies number of participants who were evaluable for this OM.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine + Oral AD | Oral AD+ Intranasal Placebo
Number analyzed (Participants) | 61 | 58
Units on a scale | 1.7 (5.02) | 4.7 (5.48)

7. Secondary Outcome: Change From Baseline in Clinical Global Impression-Severity (CGI-S) Score at Endpoint in Participants With Stable Remission (Maintenance Phase)
Description: CGI-S provides an overall clinician-determined summary measure of the severity of the participant's illness that takes into account all available information, including knowledge of the participant's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the participant's ability to function. The CGI-S evaluates the severity of psychopathology on a scale of 0 to 7. Considering total clinical experience, a participant is assessed on severity of mental illness at the time of rating according to: 0=not assessed; 1=normal (not at all ill); 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients. The change from baseline in CGI-S score, (LOCF data) at endpoint was reported. The last post baseline observation was carried forward as the endpoint.
Time Frame: Baseline and Endpoint (Up to 92 Weeks)
Population: as for outcome 5
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Intranasal Esketamine + Oral AD | Oral AD+ Intranasal Placebo
Number analyzed (Participants) | 89 | 86
Units on a scale | 0.0 [-3 to 4] | 1.0 [-2 to 5]

8. Secondary Outcome: Change From Baseline in Clinical Global Impression-Severity Score at Endpoint in Participants With Stable Response (But Not in Stable Remission) (Maintenance Phase)
Description: as for outcome 7
Time Frame: Baseline and Endpoint (Up to 92 Weeks)
Population: as for outcome 6
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Intranasal Esketamine + Oral AD | Oral AD+ Intranasal Placebo
Number analyzed (Participants) | 62 | 58
Units on a scale | 0.0 [-2 to 4] | 1.0 [-3 to 5]

9. Secondary Outcome: Change From Baseline in Generalized Anxiety Disorder-7 Items (GAD-7) Total Score at Endpoint in Participants With Stable Remission (Maintenance Phase)
Description: GAD-7 is a brief and validated 7-item self-report assessment of overall anxiety. Participants respond to each item using a 4-point scale with response categories of 0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day. Item responses are summed to yield a total score with a range of 0 to 21, where higher scores indicate more anxiety. The recall period is 2 weeks. The severity of the GAD-7 is categorized as follows: None (0-4), Mild (5-9), Moderate (10-14) and Severe (15 -21). Item responses are summed to yield a total score (range of 0 to 21), with higher scores indicating more anxiety. The change from baseline in GAD-7 total score, (LOCF data), at endpoint was reported. The last post baseline observation was carried forward as the endpoint.
Time Frame: Baseline and Endpoint (Up to 92 Weeks)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine + Oral AD | Oral AD+ Intranasal Placebo
Number analyzed (Participants) | 89 | 86
Units on a scale | 2.2 (4.45) | 4.0 (5.93)

10. Secondary Outcome: Change From Baseline in Generalized Anxiety Disorder-7 Items Total Score at Endpoint in Participants With Stable Response (But Not in Stable Remission) (Maintenance Phase)
Description: as for outcome 9
Time Frame: Baseline and Endpoint (Up to 92 Weeks)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine + Oral AD | Oral AD+ Intranasal Placebo
Number analyzed (Participants) | 61 | 58
Units on a scale | 1.4 (3.76) | 2.6 (4.26)

11. Secondary Outcome: Change From Baseline in EuroQol-5 Dimension-5 Level (EQ-5D-5L) Sum Score at Endpoint in Participants With Stable Remission (Maintenance Phase)
Description: EQ-5D-5L consists of EQ-5D-5L descriptive system and EQ visual analogue scale (EQ VAS). EQ-5D-5L descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each has 5 levels of perceived problems (1-no problem, 2-slight problems, 3-moderate problems, 4-severe problems, 5-extreme problems). Participant selects answer for each of 5 dimensions considering response that best matches his/her health "today". Responses were used to generate a Health Status Index (HSI). HSI ranges from 0 (dead) to 1.00 (full health). EQ VAS self-rating records the respondent's own assessment of his/her overall health status at time of completion, on a scale of 0 (worst health you can imagine) to 100 (best health you can imagine). Sum score ranges from 0 to 100 where, sum score = (sum of the scores from the 5 dimensions minus 5) *5. Higher score indicates worst health state.
Time Frame: Baseline and Endpoint (Up to 92 Weeks)
Population: Full (stable remitters) analysis set included all randomized participants who were in stable remission at the end of optimization phase and received at least 1 dose of intranasal study drug and 1 dose of oral AD during MA phase. Here 'N' (overall number of participants analyzed) signifies number of participants who were evaluable for this OM.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine + Oral AD | Oral AD+ Intranasal Placebo
Number analyzed (Participants) | 88 | 86
Units on a scale | 7.5 (11.87) | 10.9 (14.74)

12. Secondary Outcome: Change From Baseline in EQ Visual Analogue Scale Score at Endpoint in Participants With Stable Remission (Maintenance Phase)
Description: EQ-5D-5L is a 2-part instrument for use as a measure of health outcome, designed for self-completion by respondents. It consists of EQ-5D-5L descriptive system and EQ VAS. The EQ VAS self-rating records the respondent's own assessment of his or her overall health status at the time of completion, on a scale of 0 (the worst health you can imagine) to 100 (the best health you can imagine).
Time Frame: Baseline and Endpoint (Up to 92 Weeks)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine + Oral AD | Oral AD+ Intranasal Placebo
Number analyzed (Participants) | 88 | 86
Units on a scale | -10.4 (20.29) | -16.1 (21.80)

13. Secondary Outcome: Change From Baseline in EQ-5D-5L Health Status Index at Endpoint in Participants With Stable Remission (Maintenance Phase)
Description: EQ-5D-5L is a 2-part instrument for use as a measure of health outcome, designed for self-completion by respondents. It consists of EQ-5D-5L descriptive system and EQ VAS. EQ-5D-5L descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each has 5 levels of perceived problems (1-no problem, 2-slight problems, 3-moderate problems, 4-severe problems, 5-extreme problems). Participant selects answer for each of 5 dimensions considering response that best matches his/her health "today". Responses were used to generate a HSI. HSI ranges from 0 (dead) to 1.00 (full health).
Time Frame: Baseline and Endpoint (Up to 92 Weeks)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine + Oral AD | Oral AD+ Intranasal Placebo
Number analyzed (Participants) | 88 | 86
Units on a scale | -0.067 (0.1180) | -0.096 (0.1484)

14. Secondary Outcome: Change From Baseline in EuroQol-5 Dimension-5 Level Sum Score at Endpoint in Participants With Stable Response (But Not in Stable Remission) (Maintenance Phase)
Description: EQ-5D-5L consists of EQ-5D-5L descriptive system and EQ VAS. EQ-5D-5L descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each has 5 levels of perceived problems (1-no problem, 2-slight problems, 3-moderate problems, 4-severe problems, 5-extreme problems). Participant selects answer for each of 5 dimensions considering response that best matches his/her health "today". Responses were used to generate a HSI. HSI ranges from 0 (dead) to 1.00 (full health). EQ VAS self-rating records the respondent's own assessment of his/her overall health status at time of completion, on a scale of 0 (worst health you can imagine) to 100 (best health you can imagine). Sum score ranges from 0 to 100 where, sum score = (sum of the scores from the 5 dimensions minus 5) *5. Higher score indicates worst health state.
Time Frame: Baseline and Endpoint (Up to 92 Weeks)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine + Oral AD | Oral AD+ Intranasal Placebo
Number analyzed (Participants) | 61 | 58
Units on a scale | 3.0 (8.13) | 8.4 (13.55)

15. Secondary Outcome: Change From Baseline in EQ-5D-5L EQ Visual Analogue Scale Score at Endpoint in Participants With Stable Response (But Not in Stable Remission) (Maintenance Phase)
Description: as for outcome 12
Time Frame: Baseline and Endpoint (Up to 92 Weeks)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine + Oral AD | Oral AD+ Intranasal Placebo
Number analyzed (Participants) | 61 | 59
Units on a scale | -1.3 (15.55) | -13.8 (19.81)

16. Secondary Outcome: Change From Baseline in EQ-5D-5L Health Status Index at Endpoint in Participants With Stable Response (But Not in Stable Remission) (Maintenance Phase)
Description: as for outcome 13
Time Frame: Baseline and Endpoint (Up to 92 Weeks)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine + Oral AD | Oral AD+ Intranasal Placebo
Number analyzed (Participants) | 61 | 58
Units on a scale | -0.023 (0.0753) | -0.073 (0.1383)

17. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Total Score at Endpoint in Participants With Stable Remission (Maintenance Phase)
Description: The SDS is a participant-reported outcome measure and is a 5-item questionnaire used and accepted for assessment of functional impairment and associated disability. The first 3 items assess disruption of 1: work/school 2: social life 3: family life/home responsibilities using a 0-10 rating scale. It also has one item on days lost from school or work and one item on days when underproductive. The score for the first 3 items are summed to create a total score of 0-30 where a higher score indicates greater impairment. The recall period is 7 days. Scores <= 4 for each item and <= 12 for the total score are considered response. Scores <= 2 for each item and <= 6 for the total score are considered remission. The change from baseline in SDS total Score, (LOCF data), at endpoint was reported. The last post baseline observation was carried forward as the endpoint.
Time Frame: Baseline and Endpoint (Up to 92 Weeks)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine + Oral AD | Oral AD+ Intranasal Placebo
Number analyzed (Participants) | 82 | 77
Units on a scale | 4.7 (7.34) | 7.2 (10.44)

18. Secondary Outcome: Change From Baseline in Sheehan Disability Total Score at Endpoint in Participants With Stable Response (But Not in Stable Remission) (Maintenance Phase)
Description: as for outcome 17
Time Frame: Baseline and Endpoint (Up to 92 Weeks)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine + Oral AD | Oral AD+ Intranasal Placebo
Number analyzed (Participants) | 58 | 53
Units on a scale | 2.2 (6.63) | 6.8 (7.64)

ADVERSE EVENTS:
Time Frame: Up to 2 years
Description: Safety analysis set included all participants who received at least 1 dose of intranasal study medication or 1 dose of oral antidepressant in respective phase (Induction, Optimization, Maintenance). Follow-up analysis set included all participants who entered the follow-up phase.
Groups:
- IND: Intranasal Esketamine + Oral AD: Open-label induction (IND) phase (direct-entry participants only): received 56 milligram (mg) or 84 mg intranasal esketamine solution twice weekly with open-label oral antidepressant (AD) (one of: duloxetine/escitalopram/sertraline/venlafaxine extended release [XR]), once daily for 4 weeks.
- OP: Intranasal Esketamine + Oral AD: Optimization (OP) phase (both direct-entry and transferred-entry participants): received 56 mg or 84 mg intranasal esketamine solution once per week for the first 4 weeks, then once per week or once every other week depending on severity of depressive symptoms with open-label oral AD (one of: duloxetine/escitalopram/sertraline/venlafaxine XR), once daily for 12 weeks.
- MA: Intranasal Esketamine + Oral AD: Maintenance (MA) phase (both direct-entry and transferred-entry participants): received 56 mg or 84 mg intranasal esketamine solution once per week for the first 4 weeks, then once per week or once every other week depending on severity of depressive symptoms with open-label oral AD (one of: duloxetine/escitalopram/sertraline/venlafaxine XR), once daily until relapse or study termination.
- MA: Oral AD + Intranasal Placebo: Maintenance phase (transferred-entry participants): received intranasal esketamine matching placebo solution once per week for the first 4 weeks, then once per week or once every other week depending on severity of depressive symptoms with open-label oral AD (one of: duloxetine/escitalopram/sertraline/venlafaxine XR), until relapse or study termination.
- FU: Intranasal Esketamine + Oral AD: Participants (who were non-responders in IND phase and who were in OP and MA phase at study termination) who received at least 1 dose of 56 mg or 84 mg intranasal esketamine participated in the follow-up (FU) phase. No intranasal esketamine was administered during FU phase. Participants received oral AD for 2 weeks of the follow-up phase unless it was determined to not be clinically appropriate.
- FU: Oral AD + Intranasal Placebo: Participants (who were non-responders in IND phase and who were in OP and MA phase at study termination) who received intranasal esketamine matching placebo with oral AD participated in the FU phase. Participants received oral AD for at least the 2 weeks of the follow-up phase unless it was determined to not be clinically appropriate.
- OP_TEP: Oral AD + Intranasal Placebo: OP phase (transferred-entry participants [TEP]): received intranasal esketamine matching placebo solution once per week for the first 4 weeks, then once per week or once every other week depending on severity of depressive symptoms with open-label oral AD (one of: duloxetine/escitalopram/sertraline/venlafaxine XR), once daily for 12 weeks.
- MA_TEP: Oral AD + Intranasal Placebo: Maintenance phase (transferred-entry participants): Participants were randomized (at the end of optimization phase) to intranasal esketamine matching placebo solution once per week for the first 4 weeks, then once per week or once every other week depending on severity of depressive symptoms with open-label oral AD (one of: duloxetine/escitalopram/sertraline/venlafaxine XR).
Arm/Group | IND: Intranasal Esketamine + Oral AD | OP: Intranasal Esketamine + Oral AD | MA: Intranasal Esketamine + Oral AD | MA: Oral AD + Intranasal Placebo | FU: Intranasal Esketamine + Oral AD | FU: Oral AD + Intranasal Placebo | OP_TEP: Oral AD + Intranasal Placebo | MA_TEP: Oral AD + Intranasal Placebo
All-Cause Mortality (participants affected / at risk) | 0/437 | 0/455 | 0/152 | 0/145 | 0/481 | 0/64 | 0/86 | 0/54
Serious Adverse Events (participants affected / at risk) | 13/437 | 11/455 | 4/152 | 1/145 | 3/481 | 0/64 | 0/86 | 1/54
Other Adverse Events (participants affected / at risk) | 306/437 | 279/455 | 114/152 | 45/145 | 14/481 | 1/64 | 40/86 | 37/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IND: Intranasal Esketamine + Oral AD (N=437) | OP: Intranasal Esketamine + Oral AD (N=455) | MA: Intranasal Esketamine + Oral AD (N=152) | MA: Oral AD + Intranasal Placebo (N=145) | FU: Intranasal Esketamine + Oral AD (N=481) | FU: Oral AD + Intranasal Placebo (N=64) | OP_TEP: Oral AD + Intranasal Placebo (N=86) | MA_TEP: Oral AD + Intranasal Placebo (N=54)
Sinus Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anal Fissure (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chest Pain (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hypothermia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Autonomic Nervous System Imbalance (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lacunar Stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sedation (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Simple Partial Seizures (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ectopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 3 | 1 | 2 | 1 | 1 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Major Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mania (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Panic Attack (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Suicidal Ideation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertensive Crisis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IND: Intranasal Esketamine + Oral AD (N=437) | OP: Intranasal Esketamine + Oral AD (N=455) | MA: Intranasal Esketamine + Oral AD (N=152) | MA: Oral AD + Intranasal Placebo (N=145) | FU: Intranasal Esketamine + Oral AD (N=481) | FU: Oral AD + Intranasal Placebo (N=64) | OP_TEP: Oral AD + Intranasal Placebo (N=86) | MA_TEP: Oral AD + Intranasal Placebo (N=54)
Vertigo (Ear and labyrinth disorders) | 99 | 91 | 38 | 8 | 2 | 0 | 0 | 0
Diplopia (Eye disorders) | 16 | 10 | 9 | 0 | 0 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 45 | 30 | 24 | 1 | 0 | 0 | 0 | 0
Hypoaesthesia Oral (Gastrointestinal disorders) | 32 | 34 | 20 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 94 | 48 | 25 | 1 | 2 | 1 | 0 | 3
Paraesthesia Oral (Gastrointestinal disorders) | 16 | 13 | 8 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 29 | 17 | 10 | 1 | 0 | 0 | 0 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 5 | 22 | 11 | 12 | 1 | 0 | 0 | 13
Blood Pressure Increased (Investigations) | 34 | 26 | 10 | 5 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 97 | 61 | 31 | 7 | 0 | 1 | 6 | 0
Dizziness Postural (Nervous system disorders) | 33 | 26 | 10 | 3 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 90 | 79 | 41 | 10 | 0 | 0 | 8 | 8
Headache (Nervous system disorders) | 60 | 57 | 27 | 14 | 8 | 0 | 16 | 12
Hypoaesthesia (Nervous system disorders) | 30 | 24 | 9 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 48 | 23 | 11 | 0 | 0 | 0 | 0 | 0
Sedation (Nervous system disorders) | 43 | 19 | 10 | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 65 | 63 | 32 | 3 | 0 | 0 | 5 | 4
Anxiety (Psychiatric disorders) | 31 | 11 | 12 | 5 | 2 | 0 | 5 | 0
Confusional State (Psychiatric disorders) | 13 | 9 | 9 | 0 | 0 | 0 | 0 | 0
Dissociation (Psychiatric disorders) | 82 | 73 | 35 | 0 | 0 | 0 | 0 | 0
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 29 | 26 | 11 | 4 | 0 | 0 | 0 | 0
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 26 | 16 | 8 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2017-04-04): https://cdn.clinicaltrials.gov/large-docs/68/NCT02493868/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-16): https://cdn.clinicaltrials.gov/large-docs/68/NCT02493868/SAP_001.pdf